CLINICAL TRIAL: NCT03369418
Title: The Effect of Cranial Electrotherapy Stimulation on Emotional and Cellular Wellbeing
Brief Title: Effectiveness of CES on Emotional and Cellular Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Kirsten Tillisch, MD, MD, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-001639
Record Dates: First submitted 2016-05-19; First posted 2017-12-12 (Actual); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: devices were masked at supplier and unblinded at end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active (Active Comparator): Subjects will be given an Alpha-Stim active device for daily treatment. The electrodes attached to the device will be active. The device frequency is preset to 0.5 Hz and 100 microampere and treatment is one hour daily. The subjects will be instructed that the device is set to a low level so that the current is not detectable but should still be effective. The current will not be detectable in both active and sham devices in order for adequate blinding to occur.
  Interventions: Device: Alpha-Stim Active
- Inactive (Sham Comparator): Subjects will be given an Alpha-Stim inactive device for daily treatment. The electrodes attached to the device will be inactive. The device will not transmit anything when turned on because the electrodes are inactive. The frequency on the device will state 0.5 Hz and 100 microampere but it will not actually emit anything. Subjects in this group will receive "treatment" one hour daily. The subjects will be instructed that the device is set to a low level so that the current is not detectable but should still be effective. The current will not be detectable in both active and sham devices in order for adequate blinding to occur.
  Interventions: Device: Alpha-Stim Inactive

INTERVENTIONS:
Device: Alpha-Stim Active — The study device is a safe, commercially available take-home cranial electrotherapy stimulation device that applies an electrical current to a subject's head to treat anxiety, depression or insomnia
  Arms: Active
Device: Alpha-Stim Inactive — The study device given to the inactive group will be identical to the active except the electrodes attached to the device will be inactive. The device will not transmit anything when turned on because the electrodes are inactive.
  Arms: Inactive

SUMMARY:
The investigators aim to use a CES (cranial electrotherapy stimulation) intervention to improve emotional well-being by reducing symptoms of anxiety and depression and to assess for changes in markers of cellular health - specifically, telomere length and telomerase activity

DETAILED DESCRIPTION:
This study aims to test an auricular cranial electrotherapy stimulation (CES) device, Alpha-Stim, to assess for changes in markers of cellular health and emotional well-being improvement associated with anxiety and depression.

Returning Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF) Veterans have a high incidence of anxiety, depression, insomnia, post-traumatic stress disorder (PTSD) and chronic pain, leading to reductions in emotional well-being. This type of chronic emotional distress can lead to detrimental biological outcomes. We will compare as an exploratory outcome Veterans vs. non-Veterans response to Alpha-Stim treatment. At the cellular level, impairment of the telomere/telomerase system may be a result of this dysregulation, given the descriptions of shorter telomeres (a marker of cellular aging), as well as increased markers of inflammation in subjects with depression, anxiety and PTSD, compared to aged matched healthy populations. These negative cellular effects of emotional distress have not been well studied in this population and may offer significant benefit.

In one study of auricular CES using the same protocol proposed here, 115 patients with anxiety or anxiety and comorbid depression were studied over 5 weeks in a randomized, sham controlled trial, showing significant improvements in both anxiety and depression symptoms. Due to the complexity of overlapping negative affect symptoms that lead to impaired emotional well-being in Veterans, the investigators chose in this proposal to evaluate a composite measure of emotional distress (a combined anxiety and depression score) as the primary outcome. Beyond depression and anxiety, CES has been associated with reductions in insomnia and pain, both of which are also significant problems in Veterans, likely contributing to reduced emotional well-being.

Primarily all interested and appropriate study subjects will undergo a screening at the University of California, Los Angeles (UCLA) G. Oppenheimer Center for Neurobiology of Stress and Resilience (CNSR). The investigators expect to enroll and screen no less than 55 subjects in order to complete 22 evaluable subjects for analysis in each treatment group.

The Hospital Anxiety and Depression Scale (HADS) will assess symptom severity defined as normal range (0-7), mild (8-10), moderate (11-14) or severe (15-20). Subjects with impaired emotional well-being with mild to moderate anxiety and/or depression on the HADS scale will be included. Subjects with a maximum combined HADS score of 28 will be included. Subjects treated for anxiety, depression, psychiatric or mental health treatment must be on a stable regimen (pharmacological or non-pharmacological) for the past 3 months.

If eligible the study coordinator will contact them to schedule a screening visit at UCLA. During this visit, the research team will conduct baseline measurements via study questionnaires, history and physical exam, and a standardized psychiatric evaluation (MINI). Subjects meeting the inclusion criteria will have training in use of the Alpha-Stim device and will have their first 1 hour treatment. Subjects who tolerate the CES treatment will have blood drawn for biological measures and will take the device home to use daily for 8 weeks. Mid-study the subjects will come back to UCLA to complete questionnaires and have vital signs and weight measured. At the end of the 8 weeks, subjects will return to UCLA, return the device, have vital signs and weight measured, have the final blood draw, and complete a final set of questionnaires.

All in all, to complete the study, subjects will have an initial screening, mid and final study visit, pre, mid, and final study questionnaires, and blood drawn in the first and final visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Within the age range of 18-40 years old
3. Score 8-14 on either the anxiety or depression HADS scale as defined as mild (8-10) to moderate (11-14)
4. Subjects who receive anxiety, depression, psychiatric or mental health treatment (pharmacological or non-pharmacological) must be on a stable regimen for the past 3 months
5. No active suicidal ideation or psychosis (including schizophrenia and bipolar disorder)
6. No uncontrolled or progressive severe medical illness (e.g., cancer, uncontrolled diabetes mellitus, active cardiac disease)
7. No use of a pacemaker or any other implanted electrical device
8. No alcohol consumption greater than 2 units daily
9. Ability to independently complete the in-person study questionnaires and sign informed consent form (ICF) without assistance
10. Willing to comply with all study procedures and be available for the duration of the study
11. No participation in another clinical trial study

Exclusion Criteria:

1. Not a male
2. Younger than 18 years old or older than 40 years old
3. Score ≥15 on either the anxiety or depression HADS scale as defined as severe (15-20)
4. Subject who receive anxiety, depression, psychiatric or mental health treatment (pharmacological or non-pharmacological) who have not been on a stable regimen for the past 3 months
5. Active suicidal ideation or psychosis (including schizophrenia and bipolar disorder)
6. History of inpatient treatment or suicidal ideation within the last year
7. Use of a pacemaker or any other implanted electrical device
8. Unable to independently complete the in-person study questionnaires and sign ICF due to impaired cognitive function
9. Unwilling to comply with all study procedures
10. Unavailable for the duration of the study
11. Current participation in another clinical trial study
12. Any other condition that the investigator believes would jeopardize the safety or rights of the subject or would render the subject unable to comply with the study protocol or make use of acquired data non-analyzable

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-03; Primary Completion 2018-10-20 (Actual); Study Completion 2018-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Tillisch, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verhoeven JE, Revesz D, Wolkowitz OM, Penninx BW. Cellular aging in depression: Permanent imprint or reversible process?: An overview of the current evidence, mechanistic pathways, and targets for interventions. Bioessays. 2014 Oct;36(10):968-78. doi: 10.1002/bies.201400068. Epub 2014 Aug 20. PMID 25143317
- [Background] Simon NM, Smoller JW, McNamara KL, Maser RS, Zalta AK, Pollack MH, Nierenberg AA, Fava M, Wong KK. Telomere shortening and mood disorders: preliminary support for a chronic stress model of accelerated aging. Biol Psychiatry. 2006 Sep 1;60(5):432-5. doi: 10.1016/j.biopsych.2006.02.004. Epub 2006 Apr 11. PMID 16581033
- [Background] van Ockenburg SL, de Jonge P, van der Harst P, Ormel J, Rosmalen JG. Does neuroticism make you old? Prospective associations between neuroticism and leukocyte telomere length. Psychol Med. 2014 Mar;44(4):723-9. doi: 10.1017/S0033291713001657. Epub 2013 Jul 9. PMID 23834823
- [Background] Teyssier JR, Chauvet-Gelinier JC, Ragot S, Bonin B. Up-regulation of leucocytes genes implicated in telomere dysfunction and cellular senescence correlates with depression and anxiety severity scores. PLoS One. 2012;7(11):e49677. doi: 10.1371/journal.pone.0049677. Epub 2012 Nov 21. PMID 23185405
- [Background] Jergovic M, Tomicevic M, Vidovic A, Bendelja K, Savic A, Vojvoda V, Rac D, Lovric-Cavar D, Rabatic S, Jovanovic T, Sabioncello A. Telomere shortening and immune activity in war veterans with posttraumatic stress disorder. Prog Neuropsychopharmacol Biol Psychiatry. 2014 Oct 3;54:275-83. doi: 10.1016/j.pnpbp.2014.06.010. Epub 2014 Jun 28. PMID 24977331
- [Background] Barclay TH, Barclay RD. A clinical trial of cranial electrotherapy stimulation for anxiety and comorbid depression. J Affect Disord. 2014 Aug;164:171-7. doi: 10.1016/j.jad.2014.04.029. Epub 2014 Apr 21. PMID 24856571
- [Background] Kirsch DL, Nichols F. Cranial electrotherapy stimulation for treatment of anxiety, depression, and insomnia. Psychiatr Clin North Am. 2013 Mar;36(1):169-76. doi: 10.1016/j.psc.2013.01.006. PMID 23538086
- [Background] Lande RG, Gragnani C. Efficacy of cranial electric stimulation for the treatment of insomnia: a randomized pilot study. Complement Ther Med. 2013 Feb;21(1):8-13. doi: 10.1016/j.ctim.2012.11.007. Epub 2012 Dec 21. PMID 23374200
- [Background] Taylor AG, Anderson JG, Riedel SL, Lewis JE, Kinser PA, Bourguignon C. Cranial electrical stimulation improves symptoms and functional status in individuals with fibromyalgia. Pain Manag Nurs. 2013 Dec;14(4):327-335. doi: 10.1016/j.pmn.2011.07.002. Epub 2011 Oct 6. PMID 24315255
- [Background] Lee SH, Kim WY, Lee CH, Min TJ, Lee YS, Kim JH, Park YC. Effects of cranial electrotherapy stimulation on preoperative anxiety, pain and endocrine response. J Int Med Res. 2013 Dec;41(6):1788-95. doi: 10.1177/0300060513500749. PMID 24265330

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by flyers from the WLA VA Integrative Medicine Clinics and on the UCLA campus between April 2016 and August 2018.
Period: Overall Study
Arm/Group | Active | Inactive
Started | 16 | 14
Completed | 13 | 11
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Inactive | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.62 (7.29) | 27.09 (5.72) | 27.92 (6.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 7 | 5 | 12
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: HADS Questionnaire Combined Score
Description: The Hospital anxiety and depression scale (HADS) evaluates symptoms of anxiety and depression, minimum 0 and maximum 52 with higher scores indicating more symptoms. A combined score it utilized as the primary outcome measure, summing the scores for anxiety and depression.
Time Frame: After completion of the study (1 year)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active | Inactive
Number analyzed (Participants) | 13 | 11
score on a scale
  Baseline estimated means | 20.3077 (1.65) | 19.909 (1.79)
  Post treatment estimated mean | 11.1538 (1.65) | 15.4545 (1.79)
Statistical Analysis 1: Comparison: Active vs Inactive; Test type: Superiority — One tailed t-tests for independent groups were performed to test the hypothesis that active device will be superior to sham in decreasing the combined HAD score. This was accomplished by Contrast analysis within the framework of a random effects general linear mixed effects (RE GLMM) model; p = .013, t-test, 1 sided — A priori threshold for statistical significance was p<.05

2. Secondary Outcome: Telomere Length
Description: Telomere length will be determined using real time quantitative polymerase chain reaction (qPCR) methodology as described previously with minor modifications.30,31 Peripheral blood mononuclear cells (PBMC) are isolated and genomic DNA extracted. Using the standard curve method, cycle threshold (CT) values are plotted on a standard curve of human genomic DNA to estimate an ng/microliter concentration value. Telomere length values are expressed as the ratio of the estimated concentration generated by PCR of the telomere gene (T) divided by the hemoglobin single (S) copy gene = (T/S).
Time Frame: After completion of the study (1 year)
Population: 2 subjects had inadequate samples for analysis of telomere length, both in the active arm.
Measure: Mean (Standard Error); unit: T/S
Arm/Group | Active | Inactive
Number analyzed (Participants) | 11 | 11
T/S | .6945 (.03231) | .7841 (.03487)
Statistical Analysis 1: Comparison: Active vs Inactive; Test type: Superiority; p = .33, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study period (10 weeks).
Description: The protocol and description of adverse events (AE) and Serious adverse events (SAE) is also detailed in the protocol.
Arm/Group | Active | Inactive
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 2/13 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=13) | Inactive (N=11)
fatigue (General disorders) | 1 (1) | 0 (0)
ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
increased irritability (Psychiatric disorders) | 0 (0) | 1 (1)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — cough, sore throat and nasal congestion
vitamin d deficiency (Endocrine disorders) | 0 (0) | 1 (1)
headahce (Nervous system disorders) | 0 (0) | 1 (1)
panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
insomnia (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a feasibility study that failed to meet its recruitment goals. The results should be viewed with some caution given that the study did not reach its calculated goal sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT03369418/Prot_SAP_000.pdf